CLINICAL TRIAL: NCT06609018
Title: Clinical Investigation of Buttermere (LENS 271) Soft Contact Lenses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CV-23-02
Record Dates: First submitted 2024-09-20; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-02

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: Study includes a second phase (Parallel) that has no primary or secondary outcome measures.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Test Lenses, Then Control Lenses (Experimental): Participants will wear the Test Lenses in both eyes for one week and then cross over to the Control Lenses in both eyes for one week.
  Interventions: Device: Test Lenses (stenfilcon A); Device: Control Lenses (omafilcon A)
- Control Lenses, Then Test Lenses (Experimental): Participants will wear the Control Lenses in both eyes for one week and then cross over to the Test Lenses in both eyes for one week.
  Interventions: Device: Test Lenses (stenfilcon A); Device: Control Lenses (omafilcon A)

INTERVENTIONS:
Device: Test Lenses (stenfilcon A) — Daily disposable, soft contact lenses worn for one week
Device: Control Lenses (omafilcon A) — Daily disposable, soft contact lenses worn for one week

SUMMARY:
The purpose of the study is to compare clinical performance between two soft contact lenses.

DETAILED DESCRIPTION:
The purpose of this study is to compare clinical performance of two soft contact lenses in a crossover study over a period of 7 days of wear.

ELIGIBILITY:
Inclusion Criteria:

i. Age 8 to 18 years; at least half the population will be children or adolescents aged 8 to 15 years.

ii. Have experience with soft contact lens wear and able to insert and remove soft contact lenses.

iii. Parent/guardian and participant have read and understood the Participant Information Sheet.

iv. Parent/guardian and participant have read, signed and dated the Informed Consent and Assent (when applicable).

v. Best corrected visual acuity of at least 20/25 in each eye.

vi. Have normal eyes with the exception of the need for visual correction.

vii. Spectacle refraction:

* Age 8 to 12: -0.75D to -4.00D spherical equivalent, with cylinder ≤ -0.75D and maximum anisometropia of <1.00D
* Age 13-18: -0.75D to -7.00D spherical equivalent, with cylinder ≤ -0.75D and maximum anisometropia of <1.00D.

viii. Be willing and able to adhere to the instructions set in the clinical protocol and maintain the appointment schedule.

Exclusion Criteria:

i. Acute and subacute inflammation or infection of the anterior chamber of the eye.

ii. Any eye disease, injury, or abnormality that affects the cornea, conjunctiva, or eyelids.

iii. Severe insufficiency of lacrimal secretion (dry eyes).

iv. Corneal hypoesthesia (reduced corneal sensitivity), if not aphakic.

v. Any systemic disease that may affect the eye or be exaggerated by wearing contact lenses.

vi. Allergic reactions of ocular surfaces or adnexa that may be induced or exaggerated by wearing contact lenses or use of contact lens solutions.

vii. Any active corneal infection (bacterial, fungal, or viral).

viii. The patient is unable to follow lens handling and wear regimen or unable to obtain assistance to do so.

ix. Newly prescribed use of systemic or ocular medications for which contact lens wear could be contraindicated as determined by the investigator.

x. Monocular participants (only one eye with functional vision) or participants fit with only one lens.

xi. Subjects with slit lamp findings greater than grade 1 (e.g., edema, infiltrates, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival, anterior segment inflammation) as per ISO 11980:2012, any previous history or signs of a contact lens related corneal inflammatory event (past corneal ulcers), or any other ocular abnormality that may contraindicate contact lens wear at the enrolment visit.

xii. History of herpetic keratitis, ocular surgery or irregular cornea.

xiii. Enrolment of the family members of the investigator, family members of the investigator's staff, or individuals living in the households of these individuals.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Total Absolute Decentration | At the end of one week daily disposable wear, after at least three hours of wear.
  Total absolute decentration from pupil centre in mm at one-week follow-up visits after at least three hours of wear. Decentration for the eye in primary position (relaxed, looking straight ahead) will be measured on three-point scale where 0= optimal lens centration , 1 = acceptable decentration and 2= unacceptable decentration.
Contact Lens Centration | At the end of one week daily disposable wear, after at least three hours of wear.
  Contact lens centration clinical rating at one-week follow-up visits after at least three hours of wear. Centration for the eye in primary position (relaxed, looking straight ahead) will be measured on three-point scale where 0= optimal lens centration, 1 = acceptable decentration and 2= unacceptable decentration.
Contact Lens Movement | At the end of one week daily disposable wear, after at least three hours of wear.
  Contact lens movement at blink clinical rating at one-week follow-up visits after at least three hours of wear. Contact Lens Movement will be recorded:
  a) for the eye in the primary position immediately after the blink;
  b) for the recovery movement following digitally applied lower lid margin push-up with the lower lid as follows:
  (-2) = reduced movement unacceptable
  (-1) = reduced movement acceptable
  (0) = optimal movement
  (+1) = excessive movement acceptable
  (+2) = excessive movement unacceptable

CONTACTS AND LOCATIONS:
Overall Officials: Michel Guillon, PhD, Principal Investigator — Ocular Technology Group- International
Locations (1):
- Ocular Technology Group - International, London, United Kingdom